CLINICAL TRIAL: NCT06802484
Title: Comparing the Effects of Multicomponent Exercise on Cardiovascular Health and Lipid Profiles in Premenopausal and Postmenopausal Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Évora (Other)
Responsible Party: Principal Investigator, Bruno Figueira, Professor, University of Évora
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 22137
Record Dates: First submitted 2025-01-16; First posted 2025-01-31 (Actual); Last update posted 2025-01-31 (Actual); Status verified 2025-01

CONDITIONS: Menopause; Cardiovascular

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention)
- Pre-Menopausic (Experimental)
  Interventions: Other: Experimental: Pre-Menopausic
- Post- Menopausic (Experimental)
  Interventions: Other: Experimental: Post- Menopausic

INTERVENTIONS:
Other: Experimental: Pre-Menopausic — The physical exercise program, lasting for 26 weeks, was conducted with an uninterrupted weekly frequency of 3 sessions, on non-consecutive days, in the late afternoon (at 7:30 PM), each lasting 60 minutes.
  Arms: Pre-Menopausic
Other: Experimental: Post- Menopausic — The physical exercise program, lasting for 26 weeks, was conducted with an uninterrupted weekly frequency of 3 sessions, on non-consecutive days, in the late afternoon (at 7:30 PM), each lasting 60 minutes.
  Arms: Post- Menopausic

SUMMARY:
Background: The present study aimed to examine the effects of a 26-week multicomponent exercise program on lipid and lipoprotein profiles, blood pressure, and anthropometric parameters in healthy but sedentary premenopausal and postmenopausal women aged 40-60.

Method: The program, comprising resistance, balance, flexibility, and aerobic exercises, aimed to identify group-specific responses and establish the program's efficacy in mitigating cardiovascular risks. Seventy-five women were recruited, and 38 completed the intervention. Participants were categorized into premenopausal (n=18), postmenopausal (n=10), and control groups (n=10). Key measures included total cholesterol, low- and high-density lipoprotein cholesterol, triglycerides, glucose, systolic and diastolic blood pressure, and anthropometric variables. Statistical analyses employed the Shapiro-Wilk test, paired t-tests, Wilcoxon tests, and Kruskal-Wallis tests, with α=0.05.

ELIGIBILITY:
Inclusion Criteria:

* women aged between 40 and 60 years old;
* healthy, asymptomatic, and non-smoking;
* medical diagnosis favouring the engagement in physical-sporting activities;
* absence of clinical history related to alcoholism or uncontrolled metabolic disease;
* no clinical prescription for hypotensive pharmacological intake, cholesterol reduction, hormonal replacement therapy, or any other intervention capable of inducing alterations in lipid and lipoprotein metabolism; or
* abnormal blood sample results.

Exclusion Criteria:

* non-fulfilment of inclusion criteria;
* clinical history characterized by symptoms related to cardiovascular disease (CVD), including stroke (CVA) and coronary vascular disease (CVD), renal or hepatic disease, musculoskeletal disorders, or rheumatoid conditions that may impede full participation in the exercise program.

Ages: 40 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2024-05-01 (Actual); Primary Completion 2024-08-01 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Total Cholesterol | 26-week
Low-density lipoprotein Cholesterol | 26-week
High-density lipoprotein Cholesterol | 26-week
Triglycerides | 26-week
Castelli Risk Index I | 26-week
Castelli Risk Index II | 26-week
Very Low-Density Lipoprotein Cholesterol | 26-week
Glucose | 26-week
Systolic Blood Pressure | 26-week
Diastolic Blood Pressure | 26-week
Heart Rate | 26-week
Body Mass Index | 26-week
Waist Circumference | 26-week
Hip Circumference | 26-week
Waist Circumference/ Hip Circumference | 26-week

CONTACTS AND LOCATIONS:
Locations (1):
- Bruno Figueira, Evora, Portugal